CLINICAL TRIAL: NCT03240432
Title: Wireless Innovation for Seniors With Diabetes Mellitus (WISDM)
Brief Title: Wireless Innovation for Seniors With Diabetes Mellitus
Acronym: WISDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WISDM
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous Glucose Monitor group (Active Comparator): CGM group participants will be asked to use a Dexcom CGM sensor on a daily basis, inserting a new sensor as needed. Participants will be instructed to use the sensor according to FDA labeling. In addition, participants will be advised to check the blood glucose when symptoms or expectations do not match the CGM reading. Participants will have clinic visits at 10 days, 4 weeks, 8 weeks, 16 weeks, and 26 weeks.
  Interventions: Device: Dexcom CGM
- Blood Glucose Meter group (No Intervention): BGM group participants will be asked to use a study blood glucose meter with test strips for a fingerstick blood glucose check with a recommendation of 4 times a day. Participants will be permitted to check a fingerstick glucose as many times a day as they choose. Participants will have a phone visits at 10 days and clinic visits at 4 weeks, 8 weeks, 16 weeks, and 26 weeks. In addition to the in-clinic study visits, the BGM group will have blinded sensor placement visits one week prior to each of the 8, 16, and 26 week visits.

INTERVENTIONS:
Device: Dexcom CGM — CGM group will be instructed on how to utilize the CGM data for diabetes management. Participants will be encouraged to use CGM values for making diabetes management decisions and will be provided guidelines for when to confirm with a study BGM fingerstick.
  Arms: Continuous Glucose Monitor group

SUMMARY:
The primary objective of the study is to determine if CGM can reduce hypoglycemia and improve quality of life in older adults with T1D.

DETAILED DESCRIPTION:
Reducing hypoglycemia is an important aspect of management of T1D in older adults, many of whom have hypoglycemic unawareness, cognitive impairment, or both. CGM offers the opportunity to reduce hypoglycemia and its related complications such as fractures from falls and hospitalizations and improve quality of life including reducing hypoglycemic fear and diabetes distress. Despite these potential benefits, CGM is used by only a small proportion of older adults with T1D. Previous studies assessing CGM efficacy have included only a small number of adults ≥ 60 years of age, excluded patients most prone to severe hypoglycemia, focused on improving HbA1c rather than hypoglycemia, and used older generation CGM sensors. These studies are not generalizable to the population of older adults with T1D. The potential benefit of CGM in reducing hypoglycemia in the older adult population has not been well studied. The goal of this study is to assess the potential benefits and risks of CGM in older adults with T1D.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, all participants must meet the following criteria:

1. Clinical diagnosis of insulin dependent presumed autoimmune type 1 diabetes by the investigator and meeting at least one of the following criteria:

   i. Age > 6 months and < 10 years old at diagnosis OR ii. Positive pancreatic autoantibodies at any time (GAD-65, IA-2, ICA or ZnT8) or positive anti-insulin autoantibody at diagnosis only (within 10 days of starting insulin) OR iii. Presence of 2 or more of the following clinical indicators suggestive of type 1 diabetes:
   1. Age at diagnosis < 40 years
   2. Non-obese at diagnosis according to BMI (< 95th percentile pediatric and < 30 kg/m2 adult)
   3. Diabetic ketoacidosis (DKA) at any time,
   4. Plasma C-peptide level < 0.8 ng/ml (with blood glucose > 80 mg/dL if available) at any time
   5. Family history of type 1 diabetes in a first degree relative (parent, sibling, or child).
2. Age ≥60 years
3. HbA1c <10.0% at screening or within 30 days prior to screening visit (the upper limit was selected as a surrogate measure of likelihood of adherence to the protocol with the belief that those with higher HbA1c levels are generally noncompliant with diabetes management and thus not good candidates for the trial)
4. Insulin regimen involves either use of an insulin pump (a minimum of 40% of study population) or multiple daily injections of insulin (minimum of 40% of study population).
5. Participant is able to manage his/her diabetes with respect to insulin administration and glucose monitoring (which may include assistance from spouse or other caregiver)
6. Participant understands the study protocol and agrees to comply with it
7. Participant comprehends written and spoken English
8. At least 240 hours (10 out of 14 days) of sensor glucose data with appropriate number of calibrations from the blinded CGM pre-randomization phase

Exclusion Criteria:

Individuals meeting any of the following exclusion criteria at baseline will be excluded from study participation.

1. Use of unblinded CGM, outside of a research study, as part of real-time diabetes management in the last 3 months
2. At least 10% of time spent with sensor glucose levels < 54 mg/dl during the blinded CGM screening period AND a severe hypoglycemic event in the past 6 months (a severe hypoglycemic event that required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions (see section 8.1).
3. Extreme visual or hearing impairment that would impair ability to use real-time CGM assessed at screening visit
4. Known adhesive allergy or skin reaction during the blinded CGM pre-randomization phase that would preclude participation in the randomized trial
5. Plans to begin non-insulin medication for blood glucose lowering during the course of the study
6. Stage 4 or 5 renal disease or most recent GFR < 30 ml/min/m2 from local lab within the past 6 months
7. The presence of a significant medical or psychiatric condition or use of a medication that in the judgment of the investigator may affect completion of any aspect of the protocol, or is likely to be associated with life expectancy of <1 year.
8. Clinical diagnosis of dementia (cognitive impairment that is mild and not considered sufficient for diagnosis of dementia is acceptable)
9. Need for use of acetaminophen or acetaminophen-containing products on a regular basis during the 6 months of the trial (unless stipulation no longer required with use of newer generation sensors)
10. Inpatient psychiatric treatment in the past 6 months
11. Participation in an intervention study (including psychological studies) in past 6 weeks.
12. Expectation that participant will be moving out of the area of the clinical center during the next 6 months, unless the move will be to an area served by another study center.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Time spent with glucose level <70 mg/dL | 6 months (26 weeks) from baseline
  The primary outcome will be a treatment group comparison of the percentage of sensor values in the hypoglycemic range (<70 mg/dL), adjusted for the baseline values and factors used to stratify randomization in a regression model. Residual values will be examined for an approximate normal distribution. If values are highly skewed, then a transformation or non-parametric methods will be used instead. The BGM Group will be wearing a blinded CGM for one week at 3 time points in the study (in addition to baseline). For analysis, sensor data from the CGM Group will be used from these same time periods to match up with the blinded CGM placed for the BGM Group. The CGM data will be pooled across each time point of CGM data collection for the primary analysis.

SECONDARY OUTCOMES:
Change in HbA1c | 6 months (26 weeks) from baseline
  Mean ± SD values for the change in HbA1c from baseline to 26-weeks with 95% confidence intervals or percentiles appropriate to the distribution will be computed for each randomization group and compared in a regression model adjusted for baseline level and factors used to stratify randomization.
Change in QOL: Preferring Hypoglycemia Scale | 6 months (26 weeks) from baseline
  Mean ± SD values for the change in total score from baseline to 26-weeks with 95% confidence intervals or percentiles appropriate to the distribution will be reported for each randomization group, and compared in linear regression models adjusted for baseline level and factors used to stratify randomization.
Change in QOL: Blood glucose Monitoring Satisfaction Questionnaire | 6 months (26 weeks) from baseline
  Mean ± SD values for the change in total score from baseline to 26-weeks with 95% confidence intervals or percentiles appropriate to the distribution will be reported for each randomization group, and compared in linear regression models adjusted for baseline level and factors used to stratify randomization.
Change in QOL: Hypoglycemia Fear Survey | 6 months (26 weeks) from baseline
  Mean ± SD values for the change in total score from baseline to 26-weeks with 95% confidence intervals or percentiles appropriate to the distribution will be reported for each randomization group, and compared in linear regression models adjusted for baseline level and factors used to stratify randomization.
Change in QOL: Diabetes Distress Questionnaire | 6 months (26 weeks) from baseline
  Mean ± SD values for the change in total score from baseline to 26-weeks with 95% confidence intervals or percentiles appropriate to the distribution will be reported for each randomization group, and compared in linear regression models adjusted for baseline level and factors used to stratify randomization.
Change in QOL: PROMIS Measures for QOL | 6 months (26 weeks) from baseline
  Mean ± SD values for the change in total score from baseline to 26-weeks with 95% confidence intervals or percentiles appropriate to the distribution will be reported for each randomization group, and compared in linear regression models adjusted for baseline level and factors used to stratify randomization.
Change in QOL: NIH Cognitive Toolbox | 6 months (26 weeks) from baseline
  Mean ± SD values for the change in total score from baseline to 26-weeks with 95% confidence intervals or percentiles appropriate to the distribution will be reported for each randomization group, and compared in linear regression models adjusted for baseline level and factors used to stratify randomization.
Change in QOL: NIH Emotions Toolbox | 6 months (26 weeks) from baseline
  Mean ± SD values for the change in total and composite score from baseline to 26-weeks with 95% confidence intervals or percentiles appropriate to the distribution will be reported for each randomization group, and compared in linear regression models adjusted for baseline level and factors used to stratify randomization.
Time spent with glucose level <60 mg/dL | 6 months (26 weeks) from baseline
  Analyses will be similar to the primary objective.
Time spent with glucose level <54 mg/dL | 6 months (26 weeks) from baseline
  Analyses will be similar to the primary objective.

OTHER OUTCOMES:
Rate of episodes of severe hypoglycemia | baseline to 6 months (26 weeks)
  A hypoglycemic event will be defined as severe low blood sugar requiring assistance of another person due to altered or loss of consciousness. The rate of episodes will be tabulated and assessed using a regression model adjusted for baseline number of events.
Rate of episodes of diabetic ketoacidosis events | baseline to 6 months (26 weeks)
  A diabetic ketoacidosis event will be defined as hyperglycemia meeting all of the following criteria:
  * Symptoms such as polyuria, polydipsia, nausea, or vomiting;
  * Serum ketones >1.5 mmol/L or large/moderate urine ketones;
  * Either arterial blood pH <7.30 or venous pH <7.24 or serum bicarbonate <15; and
  * Treatment provided in a health care facility
  The rate of episodes of diabetic ketoacidosis will be tabulated and assessed using a regression model adjusted for baseline number of events.
Number of falls | baseline to 6 months (26 weeks)
  The number of falls and any resulting injuries will be tabulated and compared between treatment groups using a Fisher's exact test.
Number of ER visits | baseline to 6 months (26 weeks)
  The number of ER visits will be tabulated and compared between treatment groups using a Fisher's exact test.
Number of hospitalizations | baseline to 6 months (26 weeks)
  The number of hospitalizations will be tabulated and compared between treatment groups using a Fishers's exact test.
Number of device-related adverse events | baseline to 6 months (26 weeks)
  The study investigator will determine if an adverse event (severe hypoglycemic events, diabetic ketoacidosis events, falls, hospitalizations, ER visits, etc.) may have been caused by the study intervention (CGM) by any of the following:
  * Component disconnections
  * CGM sensors lasting fewer than 7 days
  * CGM tape adherence issues
  * Battery lifespan deficiency due to inadequate charging or extensive wireless communication
  * Intermittent device component disconnections/communication failures not leading to system replacement
  * Device issues clearly addressed in the user guide manual that do not require additional troubleshooting
  * Skin reactions from CGM sensor placement that don't meet criteria for AE reporting
  The number of device-related adverse events will be tabulated and compared between treatment groups using a Fisher's exact test.
Hyperglycemia: time >180 mg/dL | 6 months (26 weeks) from baseline
  Time spent >180 mg/dL will be compared between groups using the methods described above for the primary objective.
Hyperglycemia: time >250 mg/dL | 6 months (26 weeks) from baseline
  Time spent >250 mg/dL will be compared between groups using the methods described above for the primary objective.
Hyperglycemia: time >300mg/dL | 6 months (26 weeks) from baseline
  Time spent >300mg/dL will be compared between groups using the methods described above for the primary objective.
Hyperglycemia: area under the curve 180 mg/dL | 6 months (26 weeks) from baseline
  The area under the curve for 180 mg/dL will be compared between groups using the methods described above for the primary objective.
Hyperglycemia: high blood glucose index | 6 months (26 weeks) from baseline
  High blood glucose index will be compared between groups using the methods described above for the primary objective.
Time in range 70-180 mg/dL | 6 months (26 weeks) from baseline
  The time in range (70-180 mg/dL) will be compared between groups using the methods described above for the primary objective.
Mean glucose | 6 months (26 weeks) from baseline
  Mean glucose will be compared between groups using the methods described above for the primary objective.
Glycemic variability (coefficient of variation) | 6 months (26 weeks) from baseline
  Glycemic variability will be compared between groups using the methods described above for the primary objective.

CONTACTS AND LOCATIONS:
Overall Officials: Kellee Miller, Principal Investigator — Jaeb Center for Health Research
Locations (22):
- United States (22):
  - University of Southern California, Beverly Hills, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - University of Colorado - Barbara Davis Center, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Florida Hospital Diabetes Institute, Orlando, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University - Naomi Berrie Diabetes Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington Diabetes Care Center, Seattle, Washington

REFERENCES:
- [Derived] Miller KM, Kanapka LG, Rickels MR, Ahmann AJ, Aleppo G, Ang L, Bhargava A, Bode BW, Carlson A, Chaytor NS, Gannon G, Goland R, Hirsch IB, Kiblinger L, Kruger D, Kudva YC, Levy CJ, McGill JB, O'Malley G, Peters AL, Philipson LH, Philis-Tsimikas A, Pop-Busui R, Salam M, Shah VN, Thompson MJ, Vendrame F, Verdejo A, Weinstock RS, Young L, Pratley R. Benefit of Continuous Glucose Monitoring in Reducing Hypoglycemia Is Sustained Through 12 Months of Use Among Older Adults with Type 1 Diabetes. Diabetes Technol Ther. 2022 Jun;24(6):424-434. doi: 10.1089/dia.2021.0503. Epub 2022 Apr 11. PMID 35294272
- [Derived] Pratley RE, Kanapka LG, Rickels MR, Ahmann A, Aleppo G, Beck R, Bhargava A, Bode BW, Carlson A, Chaytor NS, Fox DS, Goland R, Hirsch IB, Kruger D, Kudva YC, Levy C, McGill JB, Peters A, Philipson L, Philis-Tsimikas A, Pop-Busui R, Shah VN, Thompson M, Vendrame F, Verdejo A, Weinstock RS, Young L, Miller KM; Wireless Innovation for Seniors With Diabetes Mellitus (WISDM) Study Group. Effect of Continuous Glucose Monitoring on Hypoglycemia in Older Adults With Type 1 Diabetes: A Randomized Clinical Trial. JAMA. 2020 Jun 16;323(23):2397-2406. doi: 10.1001/jama.2020.6928. PMID 32543682